CLINICAL TRIAL: NCT06529913
Title: Model of diseAses Related to Environmental Exposure to Heavy meTals, nanopaRticles and Emergent Contaminants, Using a dIgital platfOrm of Clinical and Bio-humoral Data: the Way to Susceptibility/RisK BiomArker [MATRIOSKA Study] - The Seed.
Brief Title: Environmental Exposure to Heavy Metals, Nanoparticles, and Emergent Contaminants and Risk of Allergic Diseases
Acronym: MATRIOSKA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Collaborators: University of Bologna (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 6628; PNC-PNRRDARE-PNC0000002 (Other Grant/Funding Number: Italian Ministry of University and Research)
Record Dates: First submitted 2024-07-26; First posted 2024-07-31 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Allergic Contact Dermatitis; Metal Allergy; Food Allergy; Nickel Sensitivity; Nickel; Eczema; Aluminum Allergy; Chromium; Eczema; Functional Gastrointestinal Disorders; Respiratory Injury; Pollution; Exposure; Pollution Related Respiratory Disorder; Environmental Exposure; Environment Related Disease; Environmental Illness; Oxidative Stress; Risk Reduction
Keywords: Metal Allergy; Nanoparticles; Emergent contaminants; Nickel; Aluminium; Copper; Chromium; Cobalt; Palladium; Titanium; Allergic Contact Dermatitis; Food Allergy; Functional Gastrointestinal Disorders; Respiratory Injury; Environmental Exposure; Patch test; Biomarkers
MeSH Terms: conditions — Dermatitis, Allergic Contact; Food Hypersensitivity; Eczema; Gastrointestinal Diseases; Environmental Illness; Risk Reduction Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Allergic contact dermatitis to metals (Experimental): Patients with allergic contact dermatitis due to metal exposure (nickel, cobalt, chromium, palladium, molybdenum, aluminium, and copper).
  Interventions: Diagnostic Test: Collection of environmental, biological, and clinical data
- Systemic allergic syndromes to metals (Experimental): Patients with systemic allergic syndrome due to metal exposure (nickel, cobalt, chromium, palladium, molybdenum, aluminium, and copper).
  Interventions: Diagnostic Test: Collection of environmental, biological, and clinical data
- Healthy volunteers (Experimental): Healthy volunteers without metal exposure (nickel, cobalt, chromium, palladium, molybdenum, aluminium, and copper).
  Interventions: Diagnostic Test: Collection of environmental, biological, and clinical data

INTERVENTIONS:
Diagnostic Test: Collection of environmental, biological, and clinical data — All enrolled patients/healthy volunteers will undergo:
  * measurement of serum and urine concentration of metals (nickel, cobalt, chromium, palladium, molybdenum, aluminium, and copper).
  * Patch test to metals.
  * Within-breath analysis of oscillometry parameters.
  * Measurement of serum zonulin.
  * Measurement of serum levels of protein oxidation products.

SUMMARY:
The goal of this clinical trial is to collect environmental, bio-humoral, and clinical data derived from patients with allergic contact dermatitis (ACD) and systemic metal allergic syndromes related to the exposure to heavy metals, nanoparticles, and emergent contaminants and from healthy subjects.

The main question it aims to answer is: are environmental, bio-humoral, and clinical data derived from patients with ACD and systemic metal allergic syndromes, related to the exposure to heavy metals, nanoparticles, and emergent contaminants, different from ones obtained by healthy subjects? Researchers will compare serum and urine concentration of heavy metals and nanoparticles, patch test to metals, within-breath analysis of oscillometry parameters, serum zonulin, and serum levels of protein oxidation products among patients with systemic allergic syndrome (1st study group), patients with ACD (2nd study group) and healthy subjects (3rd study group).

Participants will undergo:

* measurement of exposure to heavy metals and nanoparticles including nickel, cobalt, chromium, palladium, molybdenum, aluminium, and copper, through serum and urine measurement of concentration.
* Patch test to before mentioned metals.
* Within-breath analysis of oscillometry parameters.
* Measurement of serum zonulin (related to gastro-intestinal exposure).
* Measurement of serum levels of protein oxidation products (as markers of systemic oxidative stress).

DETAILED DESCRIPTION:
Heavy metals [nickel (Ni), cobalt (Co), chromium (Cr), palladium, molybdenum, aluminium, and copper] are environmental contaminants able to impact on host cells of humans and various organisms, potentially causing serious damage. These metals can be present also in form of nanoparticles.

Nanoparticles are tiny particles between 1 and 100 nanometres in size. Nanoparticles have applications in a wide range of fields, including medicine, electronics, energy, and environmental remediation. However, the potential environmental and health risks associated with nanoparticles are also focus of global research.

The research on metal allergies in exposed subjects is challenging since the exposures are common both at the workplace and outside.

Environmental exposures are important for development of allergic contact dermatitis (ACD).

ACD is a common skin disorder caused by contact with an exogenous substance that elicits a hypersensitivity response in susceptible individuals.

Among workers exposed to such irritants and allergens at work, ACD is a common occupational health problem with a significant incidence. According to the most recent scientific studies, the overall prevalence of ACD between 1996 and 2019 is estimated at 10.5 per cent.

In some individuals, the ingestion of Ni-rich foods causes systemic skin disorders (urticaria/angioedema, erythema, eczema) and extracutaneous multi-organ symptoms (heartburn, meteorism, abdominal pain, alvo, oral aphthosis, headache, respiratory disorders, recurrent infections, fibromyalgia), expressed singularly or in variable association in some particularly sensitive subjects. This clinical picture is known as Systemic Nickel Allergy Syndrome (SNAS), which occurs in approximately 20% of ACD individuals.

Researchers will collect environmental, bio-humoral, and clinical data derived from patients with ACD and systemic metal allergic syndromes related to the exposure to heavy metals, nanoparticles, and emergent contaminants, and compare with ones obtained from healthy subjects to identify susceptibility / risk factors for these diseases.

Patients with systemic allergic syndrome (1st study group) and patients with ACD (2nd study group) will undergo the measurement of exposure to heavy metals and nanoparticles including Ni, Co, Cr, palladium, molybdenum, aluminium, and copper. Furthermore, putative effect biomarkers (patch test to metals, within-breath analysis of oscillometry parameters, and serum zonulin, related to cutaneous, respiratory, and gastro-intestinal exposure, respectively, and serum levels of protein oxidation products, as markers of systemic oxidative stress) and exposure biomarkers (serum and urinary metal concentrations) will be researched in both groups. The same investigation will be conducted on healthy subjects (3rd study group).

ELIGIBILITY:
Inclusion Criteria:

* adult subjects (over 18 years of age).
* Subjects suffering from allergic contact dermatitis due to metals.
* Subjects with systemic allergic syndrome due to metals.
* Adult healthy subjects.
* Subjects able to give written informed consent.

Exclusion Criteria:

* Subjects under the age of 18years.
* Pregnant/breastfeeding women.
* Subjects suffering from chronic renal failure requiring replacement treatment.
* Subjects suffering from other systemic pathologies related to exposure to metals.
* Subjects suffering from gastrointestinal diseases such as celiac disease, chronic inflammatory intestinal diseases, tumors, other skin diseases.
* Subjects unable to express written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-05-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Serum concentration of metals | At enrollment.
  Measurement of serum concentration of heavy metals and nanoparticles including nickel, cobalt, chromium, palladium, molybdenum, aluminium, and copper.
Urinary concentration of metals | At enrollment.
  Measurement of urinary concentration of heavy metals and nanoparticles including nickel, cobalt, chromium, palladium, molybdenum, aluminium, and copper.
Patch test | At enrollment.
  Application of patch test with heavy metals including nickel, cobalt, chromium, palladium, molybdenum, aluminium, and copper.
  Patch tests will be evaluated 48h and 72h after their application and will be evaluated through a universally accepted grading system elaborated by The International Contact Dermatitis Research Group. The intensity will be assessed according to the following criteria:
  1. ± faint, non-palpable erythema;
  2. + palpable erythema;
  3. ++ strong infiltrate, numerous papules, and vesicles present strong reaction;
  4. +++ coalescing vesicles, bullae or ulceration, and an extreme erythematous reaction.
Number of subjects with altered values of respiratory system impedance | At enrollment.
  All patients and healthy volunteers will undergo oscillometry. Tidal breathing analysis with impulse oscillometry (IOS) has proven to be an informative and meaningful tool to characterize peripheral airways dysfunction.
Serum concentration of zonulin | At enrollment.
  Measurement of serum zonulin.
Serum concentration of protein oxidation products | At enrollment.
  Measurement of serum protein oxidation products as markers of systemic oxidative stress.

CONTACTS AND LOCATIONS:
Overall Officials: Angela Rizzi, MD, PhD, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (2):
- Italy (2):
  - Università di Bologna, Bologna
  - Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma

IPD SHARING:
Plan to Share IPD: No
The Researchers intend to communicate the results of the trial to participants, healthcare professionals, and other relevant groups through scientific publications and national and international conference proceedings. No individual participant data will be shared.
  All publications resulting from this research project will bear the following wording "PNC Notice DD n. 931 of 6/06/2022 - Project PNC0000002 - "DARE - Digital Lifelong Prevention".

REFERENCES:
- [Background] Rizzi A, Lo Presti E, Chini R, Gammeri L, Inchingolo R, Lohmeyer FM, Nucera E, Gangemi S. Emerging Role of Alarmins in Food Allergy: An Update on Pathophysiological Insights, Potential Use as Disease Biomarkers, and Therapeutic Implications. J Clin Med. 2023 Apr 4;12(7):2699. doi: 10.3390/jcm12072699. PMID 37048784
- [Background] Rizzi A, Chini R, Porcari S, Settanni CR, Persichetti E, Mora V, Fanali C, Leonetti A, Parrinello G, Lohmeyer FM, Inchingolo R, Mele MC, Gasbarrini A, Nucera E. Datterino Trial: A Double Blind, Randomized, Controlled, Crossover, Clinical Trial on the Use of Hydroponic Cultivated Tomato Sauce in Systemic Nickel Allergy Syndrome. J Clin Med. 2022 Sep 16;11(18):5459. doi: 10.3390/jcm11185459. PMID 36143107
- [Background] Nucera E, Rizzi A, Chini R, Giangrossi S, Lohmeyer FM, Parrinello G, Musca T, Miggiano GAD, Gasbarrini A, Inchingolo R. Diet Intervention Study through Telemedicine Assistance for Systemic Nickel Allergy Syndrome Patients during the COVID-19 Pandemic. Nutrients. 2021 Aug 23;13(8):2897. doi: 10.3390/nu13082897. PMID 34445054
- [Background] Rizzi A, Chini R, Inchingolo R, Carusi V, Pandolfi F, Gasbarrini A, Nucera E. Nickel allergy in lipid transfer protein sensitized patients: Prevalence and clinical features. Int J Immunopathol Pharmacol. 2020 Jan-Dec;34:2058738420974895. doi: 10.1177/2058738420974895. PMID 33242297
- [Background] Rizzi A, Di Rienzo A, Buonomo A, Aruanno A, Carusi V, Ricci AG, Centrone M, Mezzacappa S, Romeo L, Schiavino D, Inchingolo R, Gasbarrini A, Nucera E. Impact of nickel oral hyposensitization on quality of life in systemic nickel allergy syndrome. Int J Immunopathol Pharmacol. 2020 Jan-Dec;34:2058738420934629. doi: 10.1177/2058738420934629. PMID 32567420
- [Background] Rizzi A, Nucera E, Laterza L, Gaetani E, Valenza V, Corbo GM, Inchingolo R, Buonomo A, Schiavino D, Gasbarrini A. Irritable Bowel Syndrome and Nickel Allergy: What Is the Role of the Low Nickel Diet? J Neurogastroenterol Motil. 2017 Jan 30;23(1):101-108. doi: 10.5056/jnm16027. PMID 28049864
- [Background] Campanale M, Nucera E, Ojetti V, Cesario V, Di Rienzo TA, D'Angelo G, Pecere S, Barbaro F, Gigante G, De Pasquale T, Rizzi A, Cammarota G, Schiavino D, Franceschi F, Gasbarrini A. Nickel free-diet enhances the Helicobacter pylori eradication rate: a pilot study. Dig Dis Sci. 2014 Aug;59(8):1851-5. doi: 10.1007/s10620-014-3060-3. Epub 2014 Mar 5. PMID 24595654
- [Background] Patriarca G, Schiavino D, Pecora V, Lombardo C, Pollastrini E, Aruanno A, Sabato V, Colagiovanni A, Rizzi A, De Pasquale T, Roncallo C, Decinti M, Musumeci S, Gasbarrini G, Buonomo A, Nucera E. Food allergy and food intolerance: diagnosis and treatment. Intern Emerg Med. 2009 Feb;4(1):11-24. doi: 10.1007/s11739-008-0183-6. Epub 2008 Aug 16. PMID 18709496
- [Background] Veneroni C, Gobbi A, Pompilio PP, Dellaca R, Fasola S, La Grutta S, Leyva A, Porszasz J, Stornelli SR, Fuso L, Valach C, Breyer-Kohansal R, Breyer MK, Hartl S, Contu C, Inchingolo R, Hodgdon K, Kaminsky DA. Reference Equations for Within-Breath Respiratory Oscillometry in White Adults. Respiration. 2024;103(9):521-534. doi: 10.1159/000539532. Epub 2024 Jun 7. PMID 38843786